CLINICAL TRIAL: NCT00587639
Title: An Evaluation of Safety and Feasibility Using rTMS in Adolescents With Depression
Brief Title: An Evaluation of Safety and Feasibility Using Repetitive Transcranial Magnetic Stimulation (rTMS) in Adolescents With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Christopher A. Wall, M.D., Mayo Clinic - Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-000495
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2012-03-09 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Depression
Keywords: Adolescent; Depression; rTMS
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rTMS Treatment (Experimental): All subjects will have active rTMS treatment (10Hz, L-DLPFC - 3,000 Stimulations/treatment)
  Interventions: Device: rTMS Treatment

INTERVENTIONS:
Device: rTMS Treatment — Active rTMS treatment.
  Other Names: Neuronetics Model 2100 Therapy System

SUMMARY:
The objective of this investigation is to examine the safety and feasibility of a series of repetitive transcranial magnetic stimulation (rTMS) treatments (10 Hertz [Hz]; Left Dorsolateral Prefrontal Cortex), with a Neuronetics Model 2100 Therapy System as adjuvant treatment for depression in adolescent subjects.

DETAILED DESCRIPTION:
High frequency rTMS applied to the left dorsolateral prefrontal cortex (L-DLPFC) has been shown to have an antidepressant effect. Initial studies comparing electroconvulsive therapy (ECT) and rTMS suggest that rTMS has been as effective as ECT in treating non-psychotic depression. Given the high degree of ongoing dysfunction in depressed adolescents despite optimization of treatment with antidepressant medications, new concerns regarding suicidal thoughts and behaviors in adolescents treated with antidepressant medications, and the more interventional nature of ECT, the use of rTMS as adjuvant therapy may be of significant clinical benefit. Thus far, research using rTMS to treat depression in adolescents has been limited. The primary aim of this study is to examine the safety and feasibility of using 10 Hz rTMS applied to the left dorsolateral prefrontal cortex (L-DLPFC) as adjuvant treatment for depression in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) diagnosis of unipolar major depression without psychosis.
* Current or past history of lack of response to at least two adequate antidepressant trials selective serotonin re-uptake inhibitors (SSRI) operationally defined using the Antidepressant Treatment History Form (ATHF)
* Children's Depression Rating Scale-Revised (CDRS-R) score of 40 or higher at baseline
* At least six weeks of ongoing SSRI therapy at a stable dose.
* SSRI Medications will include:

  * Citalopram (Celexa, Cipramil, Emocal, Sepram)
  * Escitalopram oxalate (Lexapro, Cipralex, Esertia)
  * Fluoxetine (Prozac, Fontex, Seromex, Seronil, Sarafem, Fluctin (EUR))
  * Fluvoxamine maleate (Luvox, Faverin)
  * Paroxetine (Paxil, Seroxat, Aropax, Deroxat)
  * Sertraline (Zoloft, Lustral, Serlain)
* Age 13-18 years.
* Outpatient, inpatient, or partial hospitalization patients.
* Capable of providing informed assent/consent (in addition to parent/guardian consent).

Exclusion Criteria:

* Current Diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, mental retardation, pervasive developmental disorder, somatoform disorder, dissociative disorder, posttraumatic stress disorder, obsessive-compulsive disorder, eating disorders, antecedents of autism, and all personality disorders.
* Active substance dependence (except nicotine) in the past 12 months.
* Subjects with a history of head trauma, unprovoked seizure history, seizure disorder, or family history of treatment resistant epilepsy.
* Suspected pregnancy or pregnancy as confirmed by a urine pregnancy test at screening.
* History of failure to respond to ECT.
* Metal in the head (except in the mouth), implanted medication pump, cardiac pacemaker.
* Prior brain surgery.
* Risk for increased intracranial pressure such as brain tumor.
* Unable to obtain motor threshold in the subject or motor threshold too high, such that 120% MT cannot be obtained (i.e. >84% of device output).
* Significant change or increase in antidepressant medications within the last six weeks.
* Change in psychiatrist, psychologist, or therapist within the last four weeks.
* Suicide attempt within the past three months.
* Any suicide attempt or suicidal intent during the study will terminate involvement in this study.
* Subjects currently on stimulant, antipsychotic, atypical antidepressant or tricyclic antidepressant medications.
* Unstable medical or neurological conditions that may include hematological, infectious (such as Human immunodeficiency virus [HIV] positive patients) metabolic, or cardiovascular conditions that may preclude safe participation in trial.
* Subjects undergoing anticoagulant, immune suppressive and 1 or chemotherapy, or those who received any of these therapies </=3 months before enrollment in the study
* Subjects with intra-cardiac lines

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2007-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirlene M. Sampson, M.D., Principal Investigator — Mayo Clinic; Christopher A. Wall, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Rush University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - University of Texas Southwestern, Dallas, Texas

REFERENCES:
- [Result] Wall CA, Croarkin PE, Sim LA, Husain MM, Janicak PG, Kozel FA, Emslie GJ, Dowd SM, Sampson SM. Adjunctive use of repetitive transcranial magnetic stimulation in depressed adolescents: a prospective, open pilot study. J Clin Psychiatry. 2011 Sep;72(9):1263-9. doi: 10.4088/JCP.11m07003. PMID 21951987
- [Derived] Sonmez AI, Kucuker MU, Lewis CP, Kolla BP, Doruk Camsari D, Vande Voort JL, Schak KM, Kung S, Croarkin PE. Improvement in hypersomnia with high frequency repetitive transcranial magnetic stimulation in depressed adolescents: Preliminary evidence from an open-label study. Prog Neuropsychopharmacol Biol Psychiatry. 2020 Mar 8;97:109763. doi: 10.1016/j.pnpbp.2019.109763. Epub 2019 Oct 18. PMID 31634515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from clinical and community referrals at 3 participating sites. The study took place from May 2007 to October 2009.
Groups:
- Active Treatment: All subjects will have active rTMS treatment (10Hz, L-DLPFC - 3,000 Stimulations/treatment)
Period: Overall Study
Arm/Group | Active Treatment
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Active Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 16.5 (1.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Status as Measured by the Children's Auditory Verbal Learning Test 2 (CAVLT-2)
Description: The Children's Auditory Verbal Learning Test 2 (CAVLT-2) is a neuropsychological test that measures auditory verbal learning and memory. This test is designed for ages 6.6-17.11 years. Scores are reported as normalized standard scores. The minimum standard score is 60 and the maximum 140; a higher score indicates a better performance.
Time Frame: Pre-treatment (baseline visit) and post treatment (approximately 6-8 weeks after baseline visit)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rTMS Treatment
Number analyzed (Participants) | 7
units on a scale | -11.3 (12.98)

2. Secondary Outcome: Mean Level of Depression at Visit 30, as Measured by the Children's Depression Rating Scale, Revised (CDRS-R)
Description: The Children's Depression Rating Scale, Revised (CDRS-R) is a validated, 17-item, clinician rating tool to assess severity of depression. Parents provide input into 14 of the items. Scores range from 0 to 60, with the following scale: not depressed (<20), borderline depressive symptoms (20-29), mild depression (30-39), moderate depression (40-59), severe depression (>/=60).
Time Frame: At study visit 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rTMS Treatment
Number analyzed (Participants) | 7
units on a scale | 33.3 (7.3)

ADVERSE EVENTS:
Time Frame: Subjects were assessed for safety over the 6-8 weeks of treatment and at the 6- month follow-up assessment.
Description: Subjects were monitored for the possibility of headaches and scalp discomfort with a visual analog scale after each treatment.
Arm/Group | Active Treatment
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=8)
Scalp Discomfort (Skin and subcutaneous tissue disorders) | 3 (5) — Scalp discomfort is an anticipated adverse event associated with rTMS treatment.

LIMITATIONS AND CAVEATS:
Limitations of the study include its open design, and small number of total participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No